CLINICAL TRIAL: NCT02390310
Title: Simplifying the Shang Ring Technique for Circumcision of Men and Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EngenderHealth (Other)
Collaborators: Weill Medical College of Cornell University (Other); Bon Sante Consulting Limited (Unknown); Kenya National AIDS & STI Control Programme (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1084493
Record Dates: First submitted 2015-02-05; First posted 2015-03-17 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: male circumcision; Shang Ring; male circumcision device; prevention; voluntary medical male circumcision (VMMC)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Anesthesia; Lidocaine; Prilocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1 - 7 Day Removal (Active Comparator): Shang Ring No Flip Technique: Removal of Shang Ring and assessment of healing 7 days after circumcision with no-flip technique.
  Interventions: Device: Shang Ring
- Phase 1 - Delayed Removal (Active Comparator): Shang Ring No Flip Technique: Removal of ring or assessment of spontaneous detachment at more than 7 days to assess occurrence and safety following circumcision with the no-flip technique.
  Interventions: Device: Shang Ring
- Phase 2 - Topical Anesthesia (Active Comparator): Comparison of Anesthesia methods for Shang Ring circumcision: Assessment of pain during and after surgery using topical anesthesia.
  Interventions: Drug: topical anesthesia (lidocaine 2.5%, prilocaine 2.5% cream)
- Phase 2 - Injectable Anesthesia (Active Comparator): Comparison of Anesthesia methods for Shang Ring circumcision: Assessment of pain during and after surgery when using injectable anesthesia.
  Interventions: Drug: injectable anesthesia (lidocaine 1%)

INTERVENTIONS:
Device: Shang Ring — Comparison of healing times at 7 day and more than 7 days after circumcision.
  Other Names: Shang Ring No Flip Technique
  Arms: Phase 1 - 7 Day Removal; Phase 1 - Delayed Removal
Drug: injectable anesthesia (lidocaine 1%) — Comparison of Anesthesia methods for Shang Ring circumcision. Comparison of pain during Shang Ring circumcision when using injectable vs. topical anesthesia.
  Arms: Phase 2 - Injectable Anesthesia
Drug: topical anesthesia (lidocaine 2.5%, prilocaine 2.5% cream) — Comparison of Anesthesia methods for Shang Ring circumcision. Comparison of pain during Shang Ring circumcision when using injectable vs. topical anesthesia.
  Arms: Phase 2 - Topical Anesthesia

SUMMARY:
This is a research study in Kenya that will examine the outcomes of participants aged 10-15 and 16 and older; and provider acceptability of the Shang Ring technique for male circumcision that would simplify use. The study will be in two phases:

Phase 1 will explore the no-flip technique that has been used in China but will be used for the first time in Africa.

Phase 2 will be a randomized trial comparing use of tropical vs. injectable anesthesia.

DETAILED DESCRIPTION:
The study, to be conducted in two phases, will examine procedural and clinical outcomes, as well as participant and provider acceptability, of adaptations of the Shang Ring technique for male circumcision that would simplify its use and increase its acceptability.

* Phase I will be non-comparative for exploration of the no-flip technique for Shang Ring circumcision (i.e. all participants will be circumcised using the no-flip Shang Ring technique). Historical data from standard Shang Ring circumcisions conducted in Africa (Kenya, Uganda and Zambia) will be used as the comparison group. Men will be randomized to removal at 7 days after circumcision vs. delayed removal, to assess occurrence and safety of spontaneous detachments following circumcision with the no-flip technique.
* Phase 2 will compare the use of topical vs. injectable anesthesia for Shang Ring circumcision. Participants will be randomized to topical vs. injectable anesthesia in a 2:1 ratio. The investigators rationalize the 2:1 randomization scheme given that the investigators will have just completed Phase I in which 200 men and boys will have been circumcised using the no-flip technique with injected anesthesia. However, given the subjectivity associated with using reported pain as the primary endpoint, the investigators believe it is critical to randomize participants in this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 years and older;
* Uncircumcised upon clinical examination;
* In good general health;
* Free of genital ulcerations or other visible signs of sexually transmitted infections upon clinical examination;
* Participant and parent or legally acceptable representative (LAR) as applicable must be able to understand study procedures and requirements of study participation;
* Freely consents to participate in the study and signs a written informed consent form if 18 years of age or greater
* Accompanied by the parent/LAR, who freely consents and signs an informed consent form for participation of the child into the study for participants less than 18 years old;
* Assent from participant less than 18 years old who understand study procedure;
* Participant must agree to return to the study site for the full schedule of follow-up visits after his circumcision (or as appropriate the Parent or LAR must agree to bring the participant);
* Participant and parent/LAR as appropriate must agree to provide the study staff with an address, phone number, or other locator information while participating in the research study.

Exclusion Criteria:

* Has a known allergy or sensitivity to lidocaine or other local anesthesia;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
* Has known bleeding/clotting disorder (e.g. hemophilia);
* Has any congenital genitourinary abnormality;
* Has an active genital infection, anatomic abnormality or other condition (e.g. diabetes or sickle cell anemia), which in the opinion of the surgeon, prevents the man from undergoing a circumcision as part of this study; or,
* Is currently participating in another biomedical research study.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Phase I: Combined rate of moderate and severe adverse events (AEs) as a measure of safety of the no-flip technique for Shang Ring circumcision in males aged 10 years and older | 42 days
  We will evaluate the rate of moderate and severe AEs (combined) following Shang Ring MC using the no-flip technique based on clinical exam findings.
Phase 2: Pain measured with the visual analogue scale (VAS) experienced during the Shang Ring circumcision procedure with topical (EMLA Cream; lidocaine 2.5% and prilocaine 2.5%) vs. injectable (1% lidocaine) anesthesia. | 42 days
  The outcome metric for the primary outcome will be maximum pain reported to have been experienced by participants during the Shang Ring circumcision, assessed using the visual analogue scale (VAS), reported immediately after completion of the Shang Ring circumcision procedure

SECONDARY OUTCOMES:
Phase I: Ease of use of the Shang Ring with the no-flip technique as measured by MC procedure and device removal times and problems encountered during MC and removal procedures | 42 days
  To evaluate ease of use with the no-flip technique we will document MC procedure and device removal times and problems encountered during MC and removal procedures
Phase I: Satisfaction of the no-flip Shang Ring among study participants | 42 days
  we will interview participants/parents/guardians to document acceptability and satisfaction with the Shang Ring circumcision, procedure and post-procedure pain, and time to return to normal activity
Phase I: Occurrence of spontaneous detachment among those participants wearing the Shang Ring for more than 7 days days after circumcision | 42 days
  we will gather data on timing of spontaneous detachment among those participants wearing the Shang Ring for more than 7 days days after circumcision
Phase I: Safety of spontaneous detachment as measured by AEs among those participants wearing the Shang Ring for more than 7 days after circumcision | 42 days
  we will gather data to document AEs among those participants wearing the Shang Ring for more than 7 days after circumcision
Phase 2: Safety of topical vs. injectable anesthesia for local anesthesia during Shang Ring circumcision as measured by rates of moderate and severe AEs (combined rates) | 42 days
  we will document rates of moderate and severe AEs among those having a Shang Ring circumcision with topical vs. injectable anesthesia
Phase 2: Satisfaction with topical vs. injectable anesthetic among study participants | 42 days
  we will interview study participants and their parents/guardians appropriate to document acceptability and satisfaction with the circumcision, the Shang Ring procedure, post-procedure pain, and time to return to normal activity between the two techniques

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Barone, DVM, MS, Principal Investigator — EngenderHealth
Locations (2):
- Kenya (2):
  - Homa Bay Level IV County Hospital, Homa Bay, Homa Bay County
  - Vipingo Health Center, Vipingo, Kilifi County

REFERENCES:
- [Derived] Al Hussein Alawamlh O, Awori QD, Barone MA, Kim SJ, Goldstein M, Li PS, Lee RK. No-flip ShangRing circumcision in 10-12 year old boys: Results from randomized clinical trials in Kenya. PLoS One. 2020 May 22;15(5):e0233150. doi: 10.1371/journal.pone.0233150. eCollection 2020. PMID 32442198
- [Derived] Awori Q, Li PS, Lee RK, Ouma D, Oundo M, Barasa M, Obura N, Mwamkita D, Simba R, Oketch J, Nyangweso N, Maina M, Kiswi N, Kirui M, Chirchir B, Goldstein M, Barone MA. Use of topical versus injectable anaesthesia for ShangRing circumcisions in men and boys in Kenya: Results from a randomized controlled trial. PLoS One. 2019 Aug 14;14(8):e0218066. doi: 10.1371/journal.pone.0218066. eCollection 2019. PMID 31412032